CLINICAL TRIAL: NCT06141005
Title: Feasibility of Bronchial Washing Fluid for Molecular Testing With Next Generation Sequencing in Patients With Non-small Cell Lung Cancer
Brief Title: Feasibility of Bronchial Washing Fluid for Molecular Testing With Next Generation Sequencing in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2310-011-132
Record Dates: First submitted 2023-11-03; First posted 2023-11-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer
Keywords: Bronchoscopy; Liquid biopsy; Lung Cancer; Next Generation Sequencing
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrathin bronchoscopy with intratumoral washing (Experimental): Each subject suspected or diagnosed of lung cancer will undergo bronchoscopic procedure for generic alteration with Next Generation Sequencing.
  Interventions: Diagnostic Test: Ultrathin bronchoscopy with intratumoral washing

INTERVENTIONS:
Diagnostic Test: Ultrathin bronchoscopy with intratumoral washing — Each subject suspected or diagnosed of lung cancer will undergo bronchoscopic procedure. First, ultrathin bronchoscope is inserted and placed within tumor under radial EBUS, virtual bronchoscopic navigation, and fluoroscopy guidance. Then, intratumoral washing is performed. Subsequently, transbronchial lung biopsy is performed under radial EBUS, virtual bronchoscopic navigation, and fluoroscopy guidance.

SUMMARY:
This is a single center, clinical trial evaluating the relevance of intratumoral washing for detection of generic alteration with Next Generation Sequencing.

DETAILED DESCRIPTION:
This is a prospective, single-arm, open-label study to assess evaluate the relevance of intratumoral washing by ultrathin bronchoscopy (outer diameter; 3mm) for detection of genetic alterations using Next Generation Sequencing in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years
* Obtained written informed consent
* No contraindication to bronchoscopy
* Subjects suspected of having lung cancer on computed tomography or diagnosed with lung cancer by histology or cytology
* Subjects planning to undergo tissue or liquid biopsy for genetic alteration with Next Generation Sequencing

Exclusion Criteria:

* Subjects who withdraw informed consent
* Subjects who are unable to undergo liquid biopsy (plasma) and tissue biopsy for genetic alteration with Next Generation Sequencing based on the investigator's judgement
* Subjects diagnosed with a cancer other than non-small cell lung cancer from the lung tissue lesion
* Subjects diagnosed with a benign lesion from the lung tissue lesion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of the detection rate of druggable genetic alteration using Next Generation Sequencing in bronchial washing fluid, tissue, and plasma across the full patient set | through study completion, an average of 1 year
  Detection rate of druggable genetic alteration is defined as the number of true positive druggable genetic alterations detected by Next Generation Sequencing, divided by the total number of attempts. Druggable mutations were defined the presence of following genetic alterations: 1) EGFR mutation, 2) KRAS G12C mutation, 3) ALK rearrangement, 4) ROS1 rearrangement, 5) BRAF V600E mutation, 6) NTRK1/2/3 gene fusion, 7) METex14 skipping mutation, 8) RET rearrangement and 9) ERBB2 (HER2) mutation. The full patient set included all enrolled subjects.

SECONDARY OUTCOMES:
The concordance rate for the detection of druggable genetic mutations among bronchial washing fluid, plasma, and tissue samples using Next Generation Sequencing in the analysis intent group | through study completion, an average of 1 year
  The concordance rate of druggable genetic alterations detected in bronchial washing fluid by Next Generation Sequencing is compared with that in plasma and tissue in the analysis intent group. Druggable mutations were defined the presence of following genetic alterations: 1) EGFR mutation, 2) KRAS G12C mutation, 3) ALK rearrangement, 4) ROS1 rearrangement, 5) BRAF V600E mutation, 6) NTRK1/2/3 gene fusion, 7) METex14 skipping mutation, 8) RET rearrangement and 9) ERBB2 (HER2) mutation. The analysis intent group consisted of the subset of subjects for whom Next Generation Sequencing testing was successfully performed with tissue samples.
Comparisons of the detection rates of representative co-occurring genetic alterations in bronchial washing, plasma, and tissue samples across the full patient set | through study completion, an average of 1 year
  Detection rate of co-occuring genetic alteration is defined as the number of true positive co-occurring genetic alterations detected by Next Generation Sequencing, divided by the total number of attempts. Co-occurring genetic alterations were defined as the presence of following GAs: 1) ATM mutation, 2) CDKN2A mutation, 3) CTNNB1 mutation, 4) FGFR1 mutation, 5) KEAP1 mutation, 6) MDM2 amplification, 7) MET amplification, 8) MYC amplification, 9) PIK3CA mutation 10) RB1 mutation, 11) STK11 mutation and 12) TP53 mutation. The full patient set included all enrolled subjects.
The incidence of adverse events associated with the bronchial washing procedure | through study completion, an average of 1 year
  The frequency and severity of adverse events resulting from bronchial washing procedures

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Seop Eom, MD, PhD, Principal Investigator — Pusan National University Hospital
Locations (1):
- Pusan National University hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: No